CLINICAL TRIAL: NCT03412214
Title: Validity of Perfusion Index to Evaluate the Level of General Anaesthesia in Children.
Acronym: PI/AAI
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, principal investigator, Assiut University
Other Study IDs: 17300155
Record Dates: First submitted 2018-01-20; First posted 2018-01-26 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Awareness, Anesthesia
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Perfusion index detected by pulse oximeter — Perfusion index detected by pulse oximeter
  Other Names: PI
Device: AAI — The AEP Monitor/2 (Danmeter A/S, Odense, Denmark), a commercialized system for depth of anesthesia monitoring, extracts the middle latency auditory evoked potentials (MLAEP) from the EEG-signal by using an autoregressive model with an exogenous input adaptive method.
  Other Names: AAI index detected by AEP monitor.

SUMMARY:
The aim of this study is to evaluate the validity of perfusion index to determine the level of anesthesia in comparison with auditory evoked potential in children undergoing tonsillectomy.

DETAILED DESCRIPTION:
The use of the perfusion index as an added monitoring tool during anesthesia provides the anesthetist with a number of benefits. It is a useful tool to forewarn the clinician of possible light planes of anesthesia, allowing for agent dose adjustment. It is a preexisting technology that is already widely available and used in most urban, regional,and rural centers, in both developed and developing countries, is noninvasive, continuous, and inexpensive.

The AEP Monitor/2 (Danmeter A/S, Odense, Denmark), a commercialized system for depth of anesthesia monitoring, extracts the middle latency auditory evoked potentials (MLAEP) from the EEG-signal by using an autoregressive model with an exogenous input adaptive method

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3-12 years
* Elective tonsillectomy due to recurrent or chronic tonsillitis

Exclusion Criteria:

* Cerebral disease
* Cardiac disease,
* Renal disease,
* Pulmonary disease
* Hepatic disease.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: ASA physical status I-II patients aged 4-12 years and scheduled for elective tonsillectomy due to recurrent or chronic tonsillitis will be included in the study. Excluded from the study will be patients with significant cardiac, renal, pulmonary or hepatic disease.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
PI | Introperative
  Perfusion index detected by pulse oximeter
AAI index | Intraoperative
  AAI index detected by AEP monitor

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdelghaffar, MD, Principal Investigator — Professor in anesthesia and intensive care
Locations (1):
- Assiut university main hospital, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel-Ghaffar HS, Abdel-Wahab AH, Roushdy MM. Using the Perfusion Index to predict changes in the depth of anesthesia in children compared with the A-line Autoregression Index: an observational study. Braz J Anesthesiol. 2024 Sep-Oct;74(5):744169. doi: 10.1016/j.bjane.2021.04.030. Epub 2021 May 12. PMID 33991553